CLINICAL TRIAL: NCT04698863
Title: Assessment of Oxygenation With Oxygen Reserve Index for Different Fresh Gas Flows in General Anesthesia Administration
Brief Title: Assessment of Oxygenation With Oxygen Reserve Index for General Anesthesia
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, Principal investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2018-221-07/11
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Hyperoxia
Keywords: General anesthesia; Oxygen reserve index; Oxygenation; Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high flow rate: After intubation, patients had fresh gas flow with 50% O2/50% air for the first 10 minutes (3/3 L/min) and 6% desflurane. Then the flow rate was set to 4 L/min for Group High flow rate.
  Interventions: Device: Oxygen reserve index
- low flow rate: After intubation, patients had fresh gas flow with 50% O2/50% air for the first 10 minutes (3/3 L/min) and 6% desflurane. Then the flow rate was set to 1 L/min for Group Low flow rate.
  Interventions: Device: Oxygen reserve index

INTERVENTIONS:
Device: Oxygen reserve index — eveluating oxygen reserve in blood

SUMMARY:
To assess oxygenation with the oxygen reserve index in desflurane anesthesia administration using low and high fresh gas flows for tympanomastoidectomy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) risk class I-II,
* Undergoing tympanomastoidectomy

Exclusion Criteria:

* Morbid obesity
* Opioid sensitivity Alcohol or drug addiction
* Chronic obstructive pulmonary disease
* Coronary artery disease,
* Congestive heart failure
* Pronounced anemia
* Have a history of liver or kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aged between 18-65 years undergoing tympanomastoidectomy surgery
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
to assess oxygenation with the oxygen reserve index (ORI) in different fresh gas flows in general anesthesia. | During the surgery procedure
  to assess oxygenation with the oxygen reserve index (ORI) in desflurane anesthesia administration using low and high fresh gas flows for tympanomastoidectomy surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No